CLINICAL TRIAL: NCT02322970
Title: Invasive Versus Non Invasive Measurement of Intracranial Pressure in Brain Injury Trial
Brief Title: Invasive Versus Non Invasive Measurement of Intracranial Pressure in Brain Injury Trial (IMPRESSIT)
Acronym: IMPRESSIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Università degli Studi di Brescia (Other)
Collaborators: Rita Bertuetti (Unknown); Chiara Robba (Unknown)
Responsible Party: Principal Investigator, Dr. Frank Rasulo, NEURO CRITICAL CARE UNIT'S CHIEF, Università degli Studi di Brescia
Other Study IDs: impr14
Record Dates: First submitted 2014-11-10; First posted 2014-12-23 (Estimated); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Intracranial Hypertension
Keywords: intracranial hypertension; tcd; non invasive; ICP
MeSH Terms: conditions — Intracranial Hypertension; Choroideremia | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intracranial Pressure monitoring: Invasive Intracranial Pressure monitoring will be compared to non invasive intracranial monitoring ( through use of transcranial Doppler ).
  Interventions: Device: transcranial Doppler

INTERVENTIONS:
Device: transcranial Doppler — Comparison of non invasive intracranial pressure (through use of transcranial Doppler ) vs invasive monitoring (through insertion of intracerebral catheters) with the purpose of comparing these two techniques in terms of specificity and sensitivity.

SUMMARY:
Investigators aim to assess sensitivity and specificity of transcranial doppler in ruling out intracranial hypertension in all patients admitted to intensive care unit for brain injury and needing Intracranial Pressure (ICP) monitoring (according to international guidelines). Non invasive ICP measurement through the use of transcranial doppler will be carried out before and after standard invasive ICP monitoring placement.

DETAILED DESCRIPTION:
As part of intensive treatment of brain injury, intracranial pressure (ICP) should be controlled when the cerebral perfusion pressure (CPP) falls below 60-70 millimeters of mercury (mmHg) (depending on the cause of injury) and/or the ICP is greater than 20 mmHg. Intracranial hypertension (ICHP) occurs in approximately 30-40% of all patients with severe traumatic brain injury and it is not infrequent in patients with non traumatic brain injury, such as subarachnoid hemorrhage (SAH), spontaneous intracerebral hemorrhage (SICH), and ischemic stroke (IS), and the presence of ICHP and inadequate CPP has been correlated to poor outcome. Therefore, measures to monitor ICP and CPP should be instituted as soon as possible in patients with severe brain injury. Currently, available methods for ICP monitoring include epidural, subdural, subarachnoid, parenchymal, and ventricular locations. Historically, ventricular ICP catheter has been used as the reference standard and the preferred technique when possible. It is the most accurate, and reliable method of monitoring ICP. Subarachnoid, subdural, and epidural monitors are less accurate. Unfortunately, all of the described methods are invasive, associated with a complication rate and are not inexpensive. For this reason, new methods have been developed in order to measure ICP non invasively. Transcranial Doppler (TCD) allows insonation of the basal cerebral arteries and the measurement of blood flow velocities in such vessels in by using a low-frequency-pulsed Doppler of 2 Mega Hertz (MHz) over the acoustic window regions. Many authors have analysed the doppler wave shape and the relation among diastolic, systolic and mean velocities in order to find a correlation with ICP and CPP. Few formulas have been described, in our study, the method introduced and tested by Schmidt et Al. in 2000 was adopted. Those authors observed a relationship among mean arterial blood pressure (ABP) diastolic flow velocity (FVd) and mean flow velocity (FVm) in the middle cerebral artery (MCA) that led them to find a formula able to yield CPP (estimated CPP: ABP x FVd / FVm + 14); once CPP is estimated, ICPtcd is easily calculated (ICP= ABP- CPP). The first aim of our study is to evaluate the sensitivity and specificity of ICPtcd, compared to invasive ICP measurement, in order to exclude elevated ICP in patients with acute brain injury such as epidural hematomas (EDH), subdural hematomas (SDH), subarachnoid hemorrhage (SAH), intraparenchymal hemorrhage (IPH), ischaemic strokes (IS), traumatic brain injury (TBI). Inclusion criteria are:

* acute brain injury requiring invasive ICP monitoring
* Age > 18 yrs.

Exclusion criteria are:

* inaccessible or poor acoustic ultrasound window;
* a cardiovascular disease causing hemodynamic variations affecting the TCD reading (severe arrhythmia, severe cardiac valvular stenosis, moderate or severe vasospasm);
* patients receiving craniotomy or had craniectomy before first time frame 1°,
* any treatment for intracranial hypertension or manipulation of arterial blood pressure between the non-invasive ICPtcd measurements and the invasive ICP (ICPi) measurement. (This is most likely to happen during time frame 1°).

All patients included will have evaluation of non-invasive ICP monitoring through use of TCD (ICPtcd), and at least three TCD Measurements will be performed and correlated with non-invasive ICP. The timing for the TCD measurements and correlations will be as follows:

* 1° measurement: will be performed before, and as close as possible, to ICP monitoring probe placement.
* 2° measurement. Immediately following ICP monitoring probe placement;
* 3° measurement: after ICP management optimization (2-3 hours after the second measurement).

The first brain CT will be performed before invasive ICP placement (this CT scan is normally performed for diagnostic purposes) and whenever it is appropriate to perform the second scan, either for a change in clinical status, or according to guidelines and clinical judgment. If possible from 8 - 12 hrs following the first scan.

ELIGIBILITY:
Inclusion Criteria:

* Brain injury (All patients with brain injury, at risk of developing intracranial hypertension, requiring invasive intracranial pressure monitoring. );
* Patients requiring invasive ICP monitoring;
* Age > 18 yrs.

Exclusion Criteria:

* inaccessible ultrasound window;
* a cardiovascular disease causing hemodynamic variations affecting the TCD reading (severe arrhythmia, severe cardiac valvular stenosis, moderate or severe vasospasm),
* Patient already with craniotomy or craniectomy before first time frame 1°,
* any treatment for intracranial hypertension or manipulation of arterial blood pressure intervening between the non-invasive ICPtcd measurements and the invasive ICP (ICPi) measurement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with brain injury, at risk of developing intracranial hypertension, requiring invasive intracranial pressure monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 490 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of ICP tcd versus invasive ICP | 6 hours
  Analysis of specificity,sensitivity, positive predictive value and negative predictive value of trans cranial doppler in ruling out ICP above 22 mmHg (defined as intracranial hypertension) in the three different time frames

SECONDARY OUTCOMES:
ROC curve ICPtcd versus ICP | 6 hours
  Identify the best fitting ROC curve for ICP tcd in identifying intracranial hypertension.
Concordance assessment between the two methods | 6 hours
  Bland and Altman test between ICP tcd and invasive ICP is run in order to evaluate the concordance between gold standard (invasive ICP) and tcd based method

CONTACTS AND LOCATIONS:
Overall Officials: Frank A Rasulo, MD, Principal Investigator — Neuro-Intensive Care, Spedali Civili Accademic Hospital, University of Brescia, Italy
Locations (1):
- Spedali Civili, Neuro Critical Care Unit., Brescia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rasulo FA, Calza S, Robba C, Taccone FS, Biasucci DG, Badenes R, Piva S, Savo D, Citerio G, Dibu JR, Curto F, Merciadri M, Gritti P, Fassini P, Park S, Lamperti M, Bouzat P, Malacarne P, Chieregato A, Bertuetti R, Aspide R, Cantoni A, McCredie V, Guadrini L, Latronico N. Transcranial Doppler as a screening test to exclude intracranial hypertension in brain-injured patients: the IMPRESSIT-2 prospective multicenter international study. Crit Care. 2022 Apr 15;26(1):110. doi: 10.1186/s13054-022-03978-2. PMID 35428353